CLINICAL TRIAL: NCT05448469
Title: Ultrasound-guided Erector Spinae Plane Block Versus Paravertebral Block for Perioperative Analgesia, a Randomized Double Blinded Controlled Trial
Brief Title: Ultrasound-guided Erector Spinae Plane Block Versus Paravertebral Block for Perioperative Analgesia in Patients Undergoing Open Splenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R 97/2022
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- general anesthesia+ bilateral US guided erector spinae plane block (Active Comparator): General anesthesia plus ultrasound guided erector spinae plane block with 20 ml bupivacaine 0.2% at T9
  Interventions: Procedure: ultrasound guided erector spinae plane block
- general anesthesia+ bilateral US guided paravertebral block (Active Comparator): General anesthesia plus bilateral US guided paravertebral block with 7 ml bupivacaine 0.2% at T8 and T10
  Interventions: Procedure: ultrasound guided paravertebral block
- general anesthesia (Active Comparator): general anesthesia plus conventional analgesia
  Interventions: Drug: conventional analgesia

INTERVENTIONS:
Procedure: ultrasound guided erector spinae plane block — patients will receive combined general anesthesia and ultrasound guided erector spinae plane block with 20 ml of bupivacaine 0.2 % at T9 level bilaterally.
  Arms: general anesthesia+ bilateral US guided erector spinae plane block
Procedure: ultrasound guided paravertebral block — patients will receive combined general anesthesia and ultrasound guided paravertebral block with 7 ml of bupivacaine 0.2 % at T8 and T10 bilaterally.
  Arms: general anesthesia+ bilateral US guided paravertebral block
Drug: conventional analgesia — patients will receive combined general anesthesia and conventional analgesia
  Arms: general anesthesia

SUMMARY:
There are very few randomized controlled trials in open splenectomy surgery, which compare paravertebral block with ESP block. The purpose of this randomized controlled trial is to compare the efficacy of ultrasound-guided paravertebral block with ESP block for perioperative analgesia in open splenectomy .

ELIGIBILITY:
Inclusion Criteria:

* patients who will be scheduled for indicated open splenectomy surgery in the supine position via left subcostal ,midline or letf subcostal with midline extention incisions
* physical status American Society of Anesthesiologists (ASA) II or III.

Exclusion Criteria:

* Patients who refuse to participate
* patients with body mass index (BMI) >35 kg/m2
* infection at the site of injection
* coagulopathy, severe thrombocytopenia <50×103
* spine deformity
* history of opioid dependence
* polytrauma patients with dorsal spine fracture
* urgent abdominal exploration for splenectomy in heamodynamically unstable patients
* history of allergy to opioids or local anesthetics
* history of allergy to opioids, or local anaesthetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | 1st 24 hour
  all patients received an IV -PCA system (Accufuser M8P, 60 mL; Woo Young Meditech Co, S.Korea). PCA was prepared with 60 mL of isotonic saline containing 60 mg morphine, and the selected system was adjusted to infuse a 1 mL bolus dose with a lockout interval of 15 minutes while the basal flow rate was switched off. Breakthrough pain was managed with 2mg morphine.

SECONDARY OUTCOMES:
total analgesic consumption | 1st 24 hour
  The total dose of rescue analgesics(morphine) required in 24 hours will be recorded.
Numerical rating scale (NRS) | 1st 24 hour
  All patients will be monitored in the postoperative period for pain by the NRS score at rest and movement at immediate postoperative (0 min), 30 min, 1, 2, 6,12, and 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt